CLINICAL TRIAL: NCT05679375
Title: Comparison Between the Analgesic Effects of Intrathecal Versus Intravenous Ketamine After Spinal Anaesthesia for Elective Caesarean Delivery :a Randomised Trial
Brief Title: IV and Intrathecal Ketamine in Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Youstina Tharwat Sedky, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Ketamine in Cesarean section
Record Dates: First submitted 2022-12-12; First posted 2023-01-11 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Cesarean Section; Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrathecal Ketamine (Active Comparator): Patients will receive intrathecal Ketamine 0.1mg/kg added to bupivacaine and morphine.
  Interventions: Drug: Intrathecal ketamine
- Intravenous ketamine (Active Comparator): Patients will receive IV Ketamine 0.25mg/kg after spinal anesthesia with bupivacaine and morphine.
  Interventions: Drug: Intravenous ketamine

INTERVENTIONS:
Drug: Intrathecal ketamine — Patients will receive intrathecal Ketamine 0.1mg/kg added to bupivacaine and morphine
  Arms: Intrathecal Ketamine
Drug: Intravenous ketamine — Patients will receive IV Ketamine 0.25mg/kg after spinal
  Arms: Intravenous ketamine

SUMMARY:
In the current study, the investigators will compare the effects of low-dose intravenous (i.v.) ketamine versus intrathecal Ketamine added to spinal anesthesia on the time to first request for analgesia and maternal pain scores and overall satisfaction in patients undergoing cesarean section.

ELIGIBILITY:
Inclusion criteria:

• Pregnant undergoing elective cesarean section

Exclusion Criteria

* Significant coexisting diseases (pregnancy-induced hypertension or diabetes)
* body mass index ≥40kg/m2, height <150cm
* Current use of pain medication including opioids
* history of substance abuse or hallucinations, cardiovascular disease, diabetes, multiple gestations
* chronic pain was excluded.
* contraindications to spinal anaesthesia,
* severely compromised fetus requiring general anesthesia and those patients who received labor analgesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Time to the first analgesic request | First Postoperative day

SECONDARY OUTCOMES:
Postoperative pain scores NRS at rest and on movement; (2, 4, 6, 12, and 24 hours) postoperative | first postoperative day

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abd El-Rahman AM, Mohamed AA, Mohamed SA, Mostafa MAM. Effect of Intrathecally Administered Ketamine, Morphine, and Their Combination Added to Bupivacaine in Patients Undergoing Major Abdominal Cancer Surgery a Randomized, Double-Blind Study. Pain Med. 2018 Mar 1;19(3):561-568. doi: 10.1093/pm/pnx105. PMID 28520955